CLINICAL TRIAL: NCT05139329
Title: Observational Registry of Ischemia Negative Chest Pain as the Presentation of Underlying Myocarditis: the ORCHESTRATE-Myocarditis Registry
Brief Title: The ORCHESTRATE-Myocarditis Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Collaborators: Kansas City Heart Rhythm Institute (Other); Texas Cardiac Arrhythmia Research Foundation (Other); Montefiore Medical Center (Other); Loma Linda University International Heart Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: KCHRF-ORCHESTRA-0008
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Myocarditis; Ischemia; Chest Pain
MeSH Terms: conditions — Myocarditis; Ischemia; Chest Pain | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with symptoms of typical/atypical chest pain: Patients will be retrospectively included based on their presenting ICD codes or symptoms of typical/atypical chest pain, and those patients with positive ischemic workup will be excluded. The patients with negative ischemic workup will be included, and through chart review these patients will be followed to further assess their continued diagnostic workup.
  Interventions: Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Imaging — To better understand the prevalance of further imaging for evaluation of myocarditis, all patients with negative workup will be included and see what number of patients undergo further CMRI, FGD-PET, or speckle tracking echocardiography. Patients will then be categorized as those with myocarditis with positive diagnosis, negative diagnosis or unknown.

SUMMARY:
A retrospective, observational study consisting of patients who presents with typical/atypical chest pain and have an ensuing negative ischemic evaluation

DETAILED DESCRIPTION:
Multicenter, retrospective, observational study consisting of patients who presents with typical/atypical chest pain to the emergency department and have an ensuing negative ischemic evaluation. Planned to review the subsequent diagnostic process in these patients, including patients with CMRI (Cardiac Magnetic Resonance Imaging), PET (Positron Emission Tomography) imaging for evaluation of myocarditis with the goal of quantifying the number of patients who go on to have a proven diagnosis of myocarditis that can explain their presenting symptoms.

ELIGIBILITY:
Inclusion criteria

1. Age >18 years
2. Patients with a presentation of typical or atypical chest pain (ICD-10 Code R07.89, R07. 9)
3. Patients with a negative ischemic workup: (including Coronary Artery Calcium Scoring/CTA, MPI, Nuclear Stress test, LHC/angiography showing anything greater than "non-obstructive CAD")

Exclusion criteria

1. Patients with any evidence of positive ischemic workup as the cause of typical/atypical chest pain (as seen on Coronary Artery Calcium Scoring/CTA, MPI, Nuclear Stress test, LHC/angiography)
2. Previously documented history of Prinzmetal angina or coronary vasospasm
3. History of prior myocardial infarction
4. History of any prior CAD with severity greater than "non-obstructive CAD" in all 3 coronary arteries
5. History of LVEF<40%
6. Previously documented history of pericarditis
7. Previously documented history of costochondritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years of age will be included. Given the retrospective nature of this study, patients will be enrolled via chart review based upon their ICD-10 codes of chest pain on ER presentation, and these patients will be followed via chart review until a diagnosis is made. Males and females with a presentation of atypical chest pain and following a negative ischemic evaluation will be enrolled if they meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 382 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with unrecognized and underlying myocarditis | 1/2014 - 1/2022
  To quantify the number of patients with unrecognized and underlying myocarditis as a presentation of typical and atypical chest pain followed by a negative ischemic workup.

SECONDARY OUTCOMES:
Association of baseline characteristics or comorbidities with myocarditis | 1/2014 - 1/2022
  Identification of underlying baseline characteristics or comorbidities that have a greater association with myocarditis presenting as typical/atypical chest pain
Morbidity/mortality | 1/2014 - 1/2022
  Assessment morbidity/mortality in this population
Diagnostic timing for imaging modalities | 1/2014 - 1/2022
  Identification of most appropriate diagnostic timing for imaging modalities such as CMRI, FDG PET, speckle tracking echocardiography to diagnose myocarditis after initial negative ischemic workup
Comparison of specific imaging modalities | 1/2014 - 1/2022
  Comparison of specific imaging modalities (CMRI vs FDG-PET vs speckle tracking echocardiography) and their diagnostic accuracy for myocarditis
Imaging parameters that provide best diagnostic accuracy | 1/2014 - 1/2022
  Identification of specific imaging parameters on CMRI or PET imaging (late gadolinium enhancement, global dissynchrony measurements, global longitudinal strain, FDG uptake, etc) provide best diagnostic accuracy
Imaging parameters that provide best outcome prediction for morbidity/mortality | 1/2014 - 1/2022
  Identification of specific imaging parameters on CMRI or PET imaging (late gadolinium enhancement, global dissynchrony measurements, global longitudinal strain, FDG uptake, etc) provide best outcome prediction for morbidity/mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (4):
- United States (4):
  - Loma Linda University International Heart Institute, Loma Linda, California
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Montefiore Medical Center, The Bronx, New York
  - Texas Cardiac Arrhythmia Institute at St. David's Medical Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heymans S, Eriksson U, Lehtonen J, Cooper LT Jr. The Quest for New Approaches in Myocarditis and Inflammatory Cardiomyopathy. J Am Coll Cardiol. 2016 Nov 29;68(21):2348-2364. doi: 10.1016/j.jacc.2016.09.937. PMID 27884253
- [Background] Caforio AL, Pankuweit S, Arbustini E, Basso C, Gimeno-Blanes J, Felix SB, Fu M, Helio T, Heymans S, Jahns R, Klingel K, Linhart A, Maisch B, McKenna W, Mogensen J, Pinto YM, Ristic A, Schultheiss HP, Seggewiss H, Tavazzi L, Thiene G, Yilmaz A, Charron P, Elliott PM; European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Current state of knowledge on aetiology, diagnosis, management, and therapy of myocarditis: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 Sep;34(33):2636-48, 2648a-2648d. doi: 10.1093/eurheartj/eht210. Epub 2013 Jul 3. PMID 23824828
- [Background] Kindermann I, Barth C, Mahfoud F, Ukena C, Lenski M, Yilmaz A, Klingel K, Kandolf R, Sechtem U, Cooper LT, Bohm M. Update on myocarditis. J Am Coll Cardiol. 2012 Feb 28;59(9):779-92. doi: 10.1016/j.jacc.2011.09.074. PMID 22361396
- [Background] Kyto V, Sipila J, Rautava P. Acute myocardial infarction or acute myocarditis? Discharge registry-based study of likelihood and associated features in hospitalised patients. BMJ Open. 2015 May 25;5(5):e007555. doi: 10.1136/bmjopen-2014-007555. PMID 26009575
- [Background] Tornvall P, Gerbaud E, Behaghel A, Chopard R, Collste O, Laraudogoitia E, Leurent G, Meneveau N, Montaudon M, Perez-David E, Sorensson P, Agewall S. Myocarditis or "true" infarction by cardiac magnetic resonance in patients with a clinical diagnosis of myocardial infarction without obstructive coronary disease: A meta-analysis of individual patient data. Atherosclerosis. 2015 Jul;241(1):87-91. doi: 10.1016/j.atherosclerosis.2015.04.816. Epub 2015 May 1. PMID 25967935
- [Background] Vago H, Szabo L, Dohy Z, Czimbalmos C, Toth A, Suhai FI, Barczi G, Gyarmathy VA, Becker D, Merkely B. Early cardiac magnetic resonance imaging in troponin-positive acute chest pain and non-obstructed coronary arteries. Heart. 2020 Jul;106(13):992-1000. doi: 10.1136/heartjnl-2019-316295. Epub 2020 May 23. PMID 32447308
- [Background] Karamitsos TD, Arvanitaki A, Karvounis H, Neubauer S, Ferreira VM. Myocardial Tissue Characterization and Fibrosis by Imaging. JACC Cardiovasc Imaging. 2020 May;13(5):1221-1234. doi: 10.1016/j.jcmg.2019.06.030. Epub 2019 Sep 18. PMID 31542534